CLINICAL TRIAL: NCT06071442
Title: A Three-Part Phase 1 Study to Evaluate the Potential Drug-Drug Interactions Between Vemircopan and Rosuvastatin, Metformin, Levonorgestrel-Ethinyl Estradiol-Containing Oral Contraceptives, and Carbamazepine in Healthy Adult Participants
Brief Title: Potential Drug Interaction Study Between Vemircopan and Rosuvastatin, Metformin, Levonorgestrel/Ethinyl Estradiol-containing Oral Contraceptives, and Carbamazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7841C00012; ALXN2050-HV-111 (Other: Alexion)
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Drug-drug interaction; Pharmacokinetic
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin; Ethinyl Estradiol-Norgestrel Combination; Carbamazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Vemircopan, Metformin and Rosuvastatin (Experimental): Participants will receive Vemircopan, Metformin and Rosuvastatin in a fixed sequence over 2 periods.
  Period 1 (8 days): Participants will receive a single dose of metformin on day 1 and a single dose of rosuvastatin on day 4.
  Period 2 (12 days): Participants will receive vemircopan twice daily from day 1 to day 11. On day 5, participants will receive metformin co-administered with vemircopan. On day 8, participants will receive rosuvastatin co-administered with vemircopan.
  There will be a washout period of at least 4 days between the dose of rosuvastatin in Period 1 and the first dose of vemircopan in Period 2.
  Interventions: Drug: Vemircopan; Drug: Rosuvastatin; Drug: Metformin
- Part 2: Vemircopan and LNG/EE-Containing OCs (Experimental): Participants will receive Vemircopan and LNG/EE-Containing OCs in a fixed sequence over 2 periods.
  Period 1 (7 days): Participants will receive a single dose of OC, consisting of LNG and EE on day 1.
  Period 2 (10 days): Participants will receive multiple doses of vemircopan from day 1 to day 9. On day 5, participants will receive a single dose of OC co-administered with vemircopan.
  There will be a washout period of at least 7 days between the dose of OC in Period 1 and the first dose of vemircopan in Period 2.
  Interventions: Drug: Vemircopan; Drug: Levonorgestrel / Ethinyl Estradiol
- Part 3: Vemircopan and Carbamazepine (Experimental): Participants will receive Vemircopan and Carbemazepine in a fixed sequence over 2 periods.
  Period 1 (4 days): Participants will receive a single oral dose of vemircopan on day 1.
  Period 2 (22 days): Participants will receive carbemazepine twice daily from day 1 to day 21. On day 19, participants will receive a single oral dose of vemircopan co-administered with carbamazepine.
  There will be a washout period of at least 4 days between the dose of vemircopan in Period 1 and the first dose of carbamazepine in Period 2.
  Interventions: Drug: Vemircopan; Drug: Carbamazepine

INTERVENTIONS:
Drug: Vemircopan — Participants will receive oral tablets of Vemircopan.
  Other Names: ALXN2050
Drug: Rosuvastatin — Participants will receive oral coated tablets of Rosuvastatin.
  Arms: Part 1: Vemircopan, Metformin and Rosuvastatin
Drug: Metformin — Participants will receive oral film-coated tablets of Metformin.
  Arms: Part 1: Vemircopan, Metformin and Rosuvastatin
Drug: Levonorgestrel / Ethinyl Estradiol — Participants will receive oral tablets of Levonorgestrel/ Ethinyl Estradiol.
  Other Names: SIMPESSE
  Arms: Part 2: Vemircopan and LNG/EE-Containing OCs
Drug: Carbamazepine — Participants will receive oral chewable tablets of Carbamazepine.
  Arms: Part 3: Vemircopan and Carbamazepine

SUMMARY:
This study will investigate the potential drug interactions between vemircopan and metformin, rosuvastatin, levonorgestrel/ ethinyl estradiol (LNG/EE)-containing oral contraceptive(s) (OCs), and carbamazepine in healthy participants.

DETAILED DESCRIPTION:
This a 3-part drug-drug interaction (DDI) study. Part 1 - Potential Drug-drug Interaction Between Vemircopan, Metformin, and Rosuvastatin, Part 2 - Potential Drug-drug Interaction Between Vemircopan and LNG/EE-Containing OCs (Female Participants Only) Part 3 - Potential Drug-drug Interaction Between Vemircopan and Carbamazepine

All the 3 parts of the study includes:

* Screening Period: 27 days (Day -28 through Day -2)
* Two Treatment Periods:

  * Part 1: Treatment Period 1 (Day -1 through Day 8) and Treatment Period 2 (Day 1 through Day 12)
  * Part 2: Treatment Period 1 (Day -1 through Day 7) and Treatment Period 2 (Day 1 through Day 10)
  * Part 3: Treatment Period 1 (Day -1 through Day 4) and Treatment Period 2 (Day 1 through Day 22)
* Follow-up/Early Discontinuation Visit: 7 (± 2) days following the last dose of study intervention

Up to 20 participants will be enrolled per study part. Participants will be enrolled in only one study part and will not be allowed to participate in more than 1 study part.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are medically healthy with no clinically significant or relevant abnormalities as determined by medical history, physical or neurological examination, vital signs, 12-lead ECG, screening clinical laboratory profiles (hematology, biochemistry, coagulation, and urinalysis), as deemed by the Investigator or designee.
* Body weight of at minimum 50 kg and body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive) at the Screening.
* Male and female participants should adhere to the protocol defined contraceptive methods.

Exclusion Criteria:

* History or presence of medical (eg, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological or other disorders) or psychiatric conditions or diseases.
* History of clinically significant hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
* History of drug or alcohol abuse within 2 years prior to first dosing
* Current tobacco users or smokers (defined as any tobacco or nicotine-containing product use within 3 months prior to first dosing).
* Donation of whole blood from 3 months prior to first dose administration, or of plasma from 30 days before first dose administration.
* Female participants who have a positive pregnancy test at Screening or Day -1, or who are lactating.
* Positive drugs of abuse, cotinine, or alcohol screen at Screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum observed plasma (peak) concentration (Cmax) of Metformin | Up to 48 hours post-dose
  Cmax for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of metformin.
Part 1: AUC from time zero to the last quantifiable concentration (AUCt) of Metformin | Up to 48 hours post-dose
  AUCt for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of metformin.
Part 1: AUC from time zero extrapolated to infinity (AUC∞) of Metformin | Up to 48 hours post-dose
  Cmax for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of metformin.
Part 1: Cmax of Rosuvastatin | Up to 96 hours post-dose
  Cmax for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of rosuvastatin.
Part 1: AUCt of Rosuvastatin | Up to 96 hours post-dose
  AUCt for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of rosuvastatin.
Part 1: AUC∞ of Rosuvastatin | Up to 96 hours post-dose
  Cmax for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of rosuvastatin.
Part 2: Cmax of LNG | Up to 120 hours post-dose
  Cmax for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of LNG.
Part 2: AUCt of LNG | Up to 120 hours post-dose
  AUCt for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of LNG.
Part 2: AUC∞ of LNG | Up to 120 hours post-dose
  Cmax for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of LNG.
Part 2: Cmax of EE | Up to 120 hours post-dose
  Cmax for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of EE.
Part 2: AUCt of EE | Up to 120 hours post-dose
  AUCt for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of EE.
Part 2: AUC∞ of EE | Up to 120 hours post-dose
  Cmax for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on the single-dose PK of EE.
Part 3: Cmax of Vemircopan | Up to 72 hours post-dose
  Cmax for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on the single-dose PK of vemircopan.
Part 3: AUCt of Vemircopan | Up to 72 hours post-dose
  AUCt for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on the single-dose PK of vemircopan.
Part 3: AUC∞ of Vemircopan | Up to 72 hours post-dose
  Cmax for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on the single-dose PK of vemircopan.

SECONDARY OUTCOMES:
Part 1: Number of participants with Treatment Emergent Adverse Events | From Screening (Day -28 to Day -2) up to follow-up Visit or early discontinuation visit (approximately 57 days)
  The safety and tolerability of multiple doses of vemircopan when co-administered with a single dose of metformin, and multiple doses of vemircopan when co-administered with a single dose of rosuvastatin will be assessed.
Part 2: Number of participants with Treatment Emergent Adverse Events | From Screening (Day -28 to Day -2) up to follow-up Visit or early discontinuation visit (approximately 54 days)
  The safety and tolerability of multiple doses of vemircopan when co-administered with a single dose of an oral contraceptive containing both LNG and EE will be assessed.
Part 3: Number of participants with Treatment Emergent Adverse Events | From Screening (Day -28 to Day -2) up to follow-up Visit or early discontinuation visit (approximately 63 days)
  The safety and tolerability of multiple doses of vemircopan when co-administered with multiple doses of carbamazepine will be assessed.
Part 1: Time corresponding to the occurrence of Cmax (tmax) of Metformin | Up to 48 hours post-dose
  tmax for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on metformin.
Part 1: Apparent terminal elimination half-life (t½) of Metformin | Up to 48 hours post-dose
  t½ for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on metformin.
Part 1: Terminal elimination rate constant (λz) of Metformin | Up to 48 hours post-dose
  λz for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on metformin.
Part 1: Volume of distribution (apparent) following extravascular administration (Vd/F) of Metformin | Up to 48 hours post-dose
  Vd/F for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on metformin.
Part 1: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of Metformin | Up to 48 hours post-dose
  CL/F for single-dose metformin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on metformin.
Part 1: tmax of Rosuvastatin | Up to 96 hours post-dose
  tmax for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on rosuvastatin.
Part 1: t½ of Rosuvastatin | Up to 96 hours post-dose
  t½ for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on rosuvastatin.
Part 1: λz of Rosuvastatin | Up to 96 hours post-dose
  λz for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on rosuvastatin.
Part 1: Vd/F of Rosuvastatin | Up to 96 hours post-dose
  Vd/F for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on rosuvastatin.
Part 1: CL/F of Rosuvastatin | Up to 96 hours post-dose
  CL/F for single-dose rosuvastatin without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on rosuvastatin.
Part 1: Cmax of Vemircopan | Period 2: Days 4, 5 and 8
  Cmax of vermircopan after multiple twice daily doses will be assessed.
Part 1: AUC during a dosing interval at steady state (AUCtau) of Vemircopan | Period 2: Days 4, 5 and 8
  AUCtau of vermircopan after multiple twice daily doses will be assessed.
Part 1: tmax of Vemircopan | Period 2: Days 4, 5 and 8
  tmax of vermircopan after multiple twice daily doses will be assessed.
Part 1: Predose concentration prior to morning dose (Ctrough) of Vemircopan | Period 2: Days 3, 4, 5 and 8
  Ctrough of vermircopan after multiple twice daily doses will be assessed.
Part 2: tmax of LNG | Up to 120 hours post-dose
  tmax for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on LNG.
Part 2: t½ of LNG | Up to 120 hours post-dose
  t½ for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on LNG.
Part 2: λz of LNG | Up to 120 hours post-dose
  λz for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on LNG.
Part 2: Vd/F of LNG | Up to 120 hours post-dose
  Vd/F for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on LNG.
Part 2: CL/F of LNG | Up to 120 hours post-dose
  CL/F for single-dose LNG without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on LNG.
Part 2: tmax of EE | Up to 120 hours post-dose
  tmax for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on EE.
Part 2: t½ of EE | Up to 120 hours post-dose
  t½ for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on EE.
Part 2: λz of EE | Up to 120 hours post-dose
  λz for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on EE.
Part 2: Vd/F of EE | Up to 120 hours post-dose
  Vd/F for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on EE.
Part 2: CL/F of EE | Up to 120 hours post-dose
  CL/F for single-dose EE without and with co-administration with vemircopan will be assessed to determine the effect of multiple doses of vemircopan on EE.
Part 2: Cmax of Vemircopan | Period 2: Days 4, and 5
  Cmax of vermircopan after multiple twice daily doses will be assessed.
Part 2: AUCtau of Vemircopan | Period 2: Days 4, and 5
  AUCtau of vermircopan after multiple twice daily doses will be assessed.
Part 2: tmax of Vemircopan | Period 2: Days 4, and 5
  tmax of vermircopan after multiple twice daily doses will be assessed.
Part 2: Ctrough of Vemircopan | Period 2: Days 3, 4, and 5
  Ctrough of vermircopan after multiple twice daily doses will be assessed.
Part 3: tmax of Vemircopan | Up to 72 hours post-dose
  tmax for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on vemircopan.
Part 3: t½ of Vemircopan | Up to 72 hours post-dose
  t½ for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on vemircopan.
Part 3: λz of Vemircopan | Up to 72 hours post-dose
  λz for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on vemircopan.
Part 3: Vd/F of Vemircopan | Up to 72 hours post-dose
  Vd/F for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on vemircopan.
Part 3: CL/F of Vemircopan | Up to 96 hours post-dose
  CL/F for single-dose vemircopan without and with co-administration with carbamazepine will be assessed to determine the effect of multiple doses of carbamazepine on vemircopan.
Part 3: Cmax of Carbamazepine | Period 2: Days 4, 18 and 19
  Cmax of carbamazepine after multiple twice daily doses will be assessed.
Part 3: AUCtau of Carbamazepine | Period 2: Days 4, 18 and 19
  AUCtau of carbamazepine after multiple twice daily doses will be assessed.
Part 3: tmax of Carbamazepine | Period 2: Days 4, 18 and 19
  tmax of carbamazepine after multiple twice daily doses will be assessed.
Part 3: Ctrough of Carbamazepine | Period 2: Days 18 and 19
  Ctrough of carbamazepine after multiple twice daily doses will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/